CLINICAL TRIAL: NCT00583180
Title: Cutaneous Sensory Function After Wound Instillation of Capsaicin During Groin Hernia Repair
Brief Title: Sensory Function After Wound Instillation of Capsaicin
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Henrik Kehlet, Rigshospitalet
Other Study IDs: 4975-2008-01
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Primary Hyperalgesia
Keywords: Primary and/or secondary hyperalgesia; hypoesthesia
MeSH Terms: conditions — Hyperalgesia; Hypesthesia | interventions — Capsaicin; ALGRX-4975

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Capsaicin treated patients
  Interventions: Drug: Capsaicin
- P: Placebo treated patients

INTERVENTIONS:
Drug: Capsaicin — instillation of sterile water or 1000 micrograms of capsaicin into the wound at the end of open groin hernia surgery in previous study.no new intervention will be performed in the current study.
  Other Names: ALGRX 4975; ADLEA
  Groups: A

SUMMARY:
The use of capsaicin as a potential analgesic drug for postoperative pain relies on the ability of capsaicin to induce membrane lysis of c-nerve fibers. In a previous randomized placebo controled blinded study of this effect we found a significant effect of capsaicin versus placebo. Before surgery all patients were examined by quantitative sensory testing to evaluate sensory function. In this study an identical sensory testing will examine if changes to the sensory function in capsaicin treated patients is identical to placebo treated patients.No new intervention will be performed

ELIGIBILITY:
Inclusion Criteria:

* Primary groin hernia planned to undergo Lichtenstein mesh repair
* Ability to use pain scales
* American Society of Anesthesiologist class I or II based upon medical history, physical examination, and screening laboratory results
* Willing to take oral pain medication (acetaminophen, ibuprofen) for the first week
* Willing to fill out a diary for four weeks following surgery.

Exclusion Criteria:

* A previous lower abdominal surgical procedure
* Bupivacaine, acetaminophen, ibuprofen, or tramadol
* A medical condition likely to alter wound healing or pain ratings
* Systolic blood pressure greater than 150 or diastolic greater than 95 mm Hg
* Contraindication to general anesthesia
* Bilateral hernia repair
* A history of drug or alcohol abuse within the past two years
* Use of antihypertensive, antidepressant, or psychotropic drug that has not been stable for 3 months
* Use of an investigational drug within 3 months or scheduled to receive an investigational drug other than ALGRX 4975 during the study period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males with primary unilateral groin hernia
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2008-01; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
changes in sensory function before and 2 years after groin hernia repair in patients with and without capsaicin instillation, evaluated by quantitative sensory testing | 2 years

SECONDARY OUTCOMES:
Frequency of chronic pain | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, M.D, Ph. D., Study Director — Rigshospitalet, Denmark
Locations (1):
- Hørshol Sygehus, Hørsholm, Denmark